CLINICAL TRIAL: NCT02787928
Title: Dose and Response of Intrathecal Hydromorphone in Patients Undergoing Cesarean Section at Virginia Commonwealth University Health System
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of reliable supply of of preservative free IV Hydromorphone for intrathecal use.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HM20005584
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Cesarean Section; Obstetric Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intrathecal Dilaudid (Experimental): This will be a prospective up/down dosage study. After obtaining informed consent, eligible participants will be part of an up/down dose titration study. This first phase of our study will be conducted using intrathecal (spinal) hydromorphone to determine an appropriate dose range for our study population. Study drug dose will initially be 40 mcg. The only deviation from the current standard of care will be that patients will be given hydromorphone intrathecally instead of morphine. The rest of the care provided will be standard of care and per current practices at VCU labor and delivery floor.
  Interventions: Drug: Intrathecal hydromorphone

INTERVENTIONS:
Drug: Intrathecal hydromorphone — Intrathecal hydromorphone will be administered in an up/down dosage fashion. A successful dose will be defined as a patient not requiring additional narcotic pain medication outside of the standard VCU order set, which includes PRN oxycodone 5 and 10 mg every 4 hours and a one time PRN 1 mg hydromorphone IV. Failure of a dose will be if patient requires additional narcotic pain medication outside of these parameters

SUMMARY:
In the United States the incidence of cesarean deliveries have increased over the last several decades and is currently approximately 30% nationwide. The anesthesia and analgesia for elective c-sections vary between institutions.

Parturients present a unique challenge for the anesthesiologist as the mother has to care not only for herself, but also for the newborn postpartum. While intrathecal opioids provide adequate pain relief, they do so at the cost of bothersome side effects for patients, such as pruritus and nausea/vomiting.

Intrathecal hydromorphone has started to be explored as a new option for intrathecal analgesia. A study done by Beatty et al. showed in a retrospective review that 40 mcg of intrathecal dilaudid was safe and effective as compared to intrathecal morphine for analgesia after cesarean delivery. Additionally they showed no difference in side effect profiles of the two medications. Mhyre et al. investigated the use of 100 mcg of intrathecal dilaudid with hyperbaric bupivacaine in varying dosages for labor analgesia. The results were inconclusive, but the dosage of hydromorphone was reported to be without adverse effects.

Virginia Commonwealth University Health Systems has successfully instituted the use of intrathecal morphine with superior analgesia but with undesired side effects, most notably pruritus. Recent drug shortages of duramorph have prompted investigators to seek alternative options for post cesarean section analgesia. The investigators are interested in determining the dose, efficacy, and side effect profile of intrathecal hydromorphone. Although our institution has never utilized intrathecal hydromorphone for our patient population, it has been studied at various other institutions where it has been found to be safe and efficacious with an acceptable side effect profile.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status classification less than or equal to 3 Elective cesarean section Able to obtain a signed consent in English Patients who are 18 years or older

Exclusion Criteria:

* ASA greater than 3 or major medical comorbidities that are not optimized Patient refusal or contraindications to neuraxial/study drugs. Allergy to study drugs Conversion to general anesthesia Any patient who does not receive any multimodal regimen (PO acetaminophen, +/- PO ibuprofen/IV ketorolac) Any patient who is taking PO/IV opioids or buprenorphine during the current pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Narcotic Pain Medication | 12 hours post administration of intrathecal hydromorphone
  Dose failure defined as requiring more than oxycodone 5 or 10 mg q 4 hours and a 1x PRN of IV hydromorphone

SECONDARY OUTCOMES:
Nausea | 4, 8, 12, 18 and 24 hours after placement of intrathecal hydromorphone
  Rated on Numerical rating scale 0 -10 and by amount of anti-emetic medication required (ondansetron)
Pruritus | 4, 8, 12, 18 and 24 hours after placement of intrathecal hydromorphone
  Rated on numerical rating scale 0 - 10, and by amount of anti-pruritic medication required (nalbuphine, benadryl)
Sedation | 4, 8, 12, 18 and 24 hours after placement of intrathecal hydromorphone
  Richmond Agitation and Sedation Score at above time points
Pain | 4, 8, 12, 18 and 24 hours after placement of intrathecal hydromorphone
  Pain score on numeric rating scale, 0 - 10 at above time points, total amount of narcotic pain medication required
Infant Outcome | up to 10 minutes
  Infant APGAR scores at 1, 5 and 10 minutes post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Shilen Thakrar, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No